CLINICAL TRIAL: NCT05228639
Title: Coronavirus Disease 2019 Surveillance in Manhiça District Southern Mozambique for a Prompt and Effective Response Against the Epidemic
Brief Title: COVID-19 Surveillance in Rural Mozambique for Prompt and Effective Response
Acronym: MozCOVID
Status: Completed | Type: Observational
Sponsor: Centro de Investigacao em Saude de Manhica (Other)
Collaborators: Barcelona Institute for Global Health (Other); Imperial College London (Other); Instituto Nacional de Saúde, Mozambique (Other Government); Instituto de Biomedina de Valencia, IBV (Unknown); World Health Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 80/CNBS/20
Record Dates: First submitted 2022-02-04; First posted 2022-02-08 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
Keywords: SARS-CoV-2 infection; Epidemiology; Diagnostic; Surveillance; Serosurvey
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Nasopharyngeal swabs to detect SARS-CoV-2, blood, feces, and saliva samples are being collect from the study participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extraordinary times require extraordinary measures. The current COVID-19 pandemic is the paradigmatic example of how infectious diseases may menace the world's health and economy, and particularly contribute to enhancing current inequities in health-related to wealth. The main goal of the proposed study is to understand the epidemiology and natural history of COVID-19 in a rural area in Southern Mozambique

DETAILED DESCRIPTION:
Although Mozambique has so far had few confirmed cases of COVID19, it is unknown if low testing rates and other factors such as the warm climatic conditions may explain the apparently low spread of the virus. The present proposal aims to rapidly gain an understanding of the epidemic curve and natural history of SARS-CoV-2 in a rural area in southern Mozambique through a series of epidemiological indicators obtained at both the health facility and community levels, so as to provide evidence-based recommendations for managing and mitigating the COVID19 epidemic. Age-specific incidence of severe COVID-19 obtained at health facilities during a period of 15 months together with seroprevalence data obtained from the community will be used to determine SARS-CoV-2 reproduction number and effects of interventions through mathematical modeling. Viral, serological, and clinical progression will be assessed in a longitudinal cohort of symptomatic SARS-CoV-2 infected individuals. Community awareness of COVID-19 and of project aims will be fostered through engagement activities among community leaders and members. COVID-19 surveillance capacities in Mozambique will be strengthened by developing SARS-CoV-2 diagnostic approaches (molecular testing and an innovative immunoassay to detect antibodies against the virus), as well as SARS-CoV-2 genome sequencing approaches to identify transmission chains. Finally, the project will pursue the creation of a bank of serum, virus materials, and data which will be open for immediate public health purposes, including the development of point-of-care diagnostic tests. This project will be coordinated by the Manhiça Health Research Centre (Mozambique) in conjunction with the Barcelona Institute for Global Health (Spain), which will lead the transfer of molecular and immunological tools to the Mozambican research center. Imperial College will provide the modeling expertise to derive metrics of transmission, and INS the expertise to conduct quality control of laboratory determinations as well as dissemination and networking with the Ministry of Health in Mozambique. Four WPs will comprise the main research tasks, including COVID-19 surveillance (WP1), Laboratory determinations (WP2), Contact tracing and community awareness (WP3), Modelling (WP4), as well as two cross-cutting WPs related to Capacity-building (WP5) and Scientific coordination, management, networking & dissemination (WP6). We expect this 21-month project will increase the level of preparedness, alertness, and response in Mozambique

ELIGIBILITY:
Inclusion Criteria The study has five components and therefore the inclusion criteria may vary from one component to another.

1. COVID-19 morbidity surveillance

   * Individuals of any age admitted to MDH or pregnant attending the Maragra health center meet the COVID-19 case definition as defined above after the project start date.
   * Resident of Manhiça DSS area
   * Written informed consent from a parent or guardian if a child, and from participant if an adult prior recruitment.
2. COVID-19 mortality surveillance • All deaths in children under the age of 5 (including stillbirths), occurring at the health facility or at the community; • In hospital adult deaths occurring at the MDH;

   • Resident of Manhiça DSS area;

   • Written informed consent from the relative of the dead person.
3. COVID-19 population-based serosurveys • Individuals of all age groups residing in Manhiça DSS surveillance area • Signed informed parental permission from a parent or guardian if a child and from participant if an adult.
4. Natural history of SARS-CoV-2 infection

   • Participants who fulfill eligibility criteria for activity a) and with laboratory-confirmed SARS-CoV-2 infection.
5. Clinical presentation and factors associated with SARS-CoV-2 • Participants who fulfill eligibility criteria for activities a) and c).

Exclusion Criteria

• Participation in an interventional clinical trial at the time of enrollment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Manhiça district has a total population of 204,357 and 47.061 households and 27.560 children under five years. Each person living within the DSS study area is issued a unique Permanent Identification number that describes the geographic localization of his/her household. Some demographic indicators in 2015 are: a birth cohort of 3,946, life expectancy at birth 51 years, neonatal, infant, and under-five mortalities are 22.5/1,000 live births, 55.8 and 99.0, respectively. Children under the age of five represent 18% (29,700) of the total population.
Sampling Method: Non-Probability Sample
Enrollment: 6494 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Age-specific positivity rate of SARS-CoV-2 infection | 15 months
  Positivity rate by age-group (0-9, 10-19, 20-29, 30-39, 40-49, 50-59, 60-69, >=70 years) of SARS-CoV-2 infection among acute respiratory syndrome individuals during 15 months
Age-specific Incidence of SARS-CoV-2 infection | 15 months
  Incidence by age-group (0-9. 10-19, 20-29, 30-39, 40-49, 50-59, 60-69, >=70 years) of SARS-CoV-2 infection among acute respiratory syndrome individuals during 15 months
Community Age-specific seroprevalence | month 5
  Seroprevalence by age-group (0-19, 20-39, 40-59, >=60 years) of IgM and IgG against SARS-CoV-2 at baseline andd after 15 months
Community Age-specific seroprevalence | month 11
  Seroprevalence by age-group (0-19, 20-39, 40-59, >=60 years) of IgM and IgG against SARS-CoV-2 at baseline andd after 15 months
Community Age-specific seroprevalence | month 14
  Seroprevalence by age-group (0-19, 20-39, 40-59, >=60 years) of IgM and IgG against SARS-CoV-2 at baseline andd after 15 months
COVID-19 associated mortality | 2 years
  Factors associated with acute COVID-19, sero-positivity and COVID-19 associated mortality

SECONDARY OUTCOMES:
PCR and antibody-negativization | up to 12 months
  Median time (weeks or months) to PCR and antibody-negativization in symptomatic PCR-confirmed acute COVID-19 individuals
Relatedness of SARS-CoV-2 genome | 15 months
  Monophyletic groups of closely related SARS-CoV-2 genome

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de investigacao em saude de Manhica, Manhiça, Mozambique